CLINICAL TRIAL: NCT01097070
Title: A Phase II Multicenter, Open-label, Randomized, Parrallel Group Study to Assess the Pharmacokinetics of Bevirimat (BVM) 100 mg Tablets Administered to HIV-1 Positive Patients for 15 Days
Brief Title: A Phase 2 Study to Assess the Pharmacokinetics of Bevirimat 100 mg Tablets Given to HIV-1 Positive Patient for 15 Days
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Myrexis Inc. (Industry)
Responsible Party: Andrew Beelen, MD., Study Director, Myriad Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Bevirimat Study 206
Record Dates: First submitted 2010-03-23; First posted 2010-04-01 (Estimated); Last update posted 2010-04-01 (Estimated); Status verified 2010-03

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — bevirimat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Bevirimat 200 mg twice daily, 15 days (Experimental)
  Interventions: Drug: Bevirimat
- Bevirimat 300 mg once daily, 15 days (Experimental)
  Interventions: Drug: Bevirimat
- Bevirimat 400 mg once daily, 15 days (Experimental)
  Interventions: Drug: Bevirimat

INTERVENTIONS:
Drug: Bevirimat
  Other Names: MPC-4326

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, and pharmacokinetics (behavior in the body) of bevirimat administered for 15 days to HIV-positive individuals.

ELIGIBILITY:
Inclusion Criteria:

* Have documentation of HIV-1 infection in their medical records (documentation of any prior plasma viremia is acceptable).
* Have a CD4+ lymphocyte count >/= 100 cells/mm3.
* Have a screening plasma HIV-1 RNA value, measured by the Roche Amplicor assay, of <400 copies/mL.
* Be receiving an ARV therapy regimen containing at least 3 drugs which has been unchanged for at least 8 weeks prior to screening, and which is to be continued through Day 15 of the study.
* Be informed of the nature of the study and provide written informed consent.
* Be legally competent and able to communicate effectively with study personnel.
* Be able and willing to comply with outpatient visits.

Exclusion Criteria:

* Presence of any acute illness within 14 days prior to study entry.
* Presence of any AIDS-related opportunistic infection (Category C according to the CDC Classification System for HIV-1 Infection, 1993 Revised Version) that is unstable in the Investigator's opinion or diagnosed in the 30 days prior to study entry.
* Patients who are, in the opinion of the Investigator, unable to comply with the dosing schedule and protocol evaluations.
* Patients with malabsorption syndromes affecting drug absorptions (e.g. Crohn's disease, chronic pancreatitis).
* Patients with systolic blood pressure < 90 mmHg or > 160 mmHg or diastolic blood pressure < 50 mmHg or > 110 mmHg.
* A history of seizures (excluding pediatric febrile seizures) or current administration of prophylactic anti-seizure medication for the indication of seizures or seizure-related conditions.
* A history of cerebrovascular accident (CVA) or transient ischemic attacks (TIA).
* Patients who have received radiation therapy or cytotoxic chemotherapeutic agents within 4 weeks prior to first dose of study drug.
* Patients who have received treatment with immunomodulating agents such as IL-2, alpha-interferon, beta-interferon, or gamma-interferon within 4 weeks prior to first dose of study drug.
* Receipt of an investigational drug or product, or participation in a drug study within a period of 30 days prior to receiving study medication.
* Bupropion-containing products require at least a 14-day washout period and will not be approved for co-administration.
* Rifampin or other rifamycin products require at least a 28-day washout period and will not be approved for coadministration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-11; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Measure bevirimat blood plasma concentrations to calculate the pharmacokinetic parameters of AUC, Cmax, Cmin, and half-life when bevirimat is administered as 2 x 100 mg tablets BID, 3 X 100 mg tablets QD, 4 X 100 mg tablets QD for 15 days | 16 days

SECONDARY OUTCOMES:
Measure bevirimat blood plasma concentrations following the administration of bevirimat 2 X 100 mg, 3 x 100 mg, or 4 x 100 mg tablets after a standardized meal. The pharmacokinetic parameters of AUC, Cmax, Cmin, and half-life will be calculated. | Day 15

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Beelen, MD, Study Director — Myrexis Inc.; Jacob P Lalezari, MD, Principal Investigator — Quest Clinical Research; Gary J Richmond, MD, PA, Principal Investigator; Melanie A Thompson, MD, Principal Investigator — AIDS Research Consortium of Atlanta; Calvin J Cohen, MD, MSc, Principal Investigator — Community Research Initiative of New England
Locations (4):
- United States (4):
  - Quest Clinical Research, San Francisco, California
  - Gary J. Richmond, MD, PA, Fort Lauderdale, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Community Research Initiative of New England, Boston, Massachusetts